CLINICAL TRIAL: NCT05858424
Title: Impact Evaluation of a Multidisciplinary End-of-treatment Day Hospital on the Quality of Life of Adolescents and Young Adults with Cancer
Brief Title: Impact of a Multidisciplinary End-of-treatment Day Hospital on the Quality of Life of Adolescents and Young Adults with Cancer
Acronym: HOPAYA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ET22000179
Record Dates: First submitted 2022-10-20; First posted 2023-05-15 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor; Lymphoma
Keywords: Survivorship; Supportive care needs; Adolescents and Young Adults; Post-treatment; Oncology; Quality of life
MeSH Terms: conditions — Lymphoma; Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a monocentric open-label clinical research with 2 parallel groups. Patients will be 1:1 randomly assigned in both groups.
  * Group A : former patients with multidisciplinary day hospitalization
  * Group B : former patients without multidisciplinary day hospitalization
Who Masked: Participant, Investigator
Masking Description: Randomization will be performed according to a minimization algorithm of the Ennov Clinical software. The ratio will be 1:1 by stratifying on the criterion: management service (CLB vs IHOPe).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A : former patients with multidisciplinary day hospitalization (Experimental): In this group, a multidisciplinary day hospitalization will be programmed after the end-of-treatment evaluation and 2 months after the end of treatment at the latest. This day hospitalization will consist at least of a psychological interview, an interview with a social worker and a medical interview.
  Interventions: Other: Multidisciplinary day hospitalization
- Group B : former patients without multidisciplinary day hospitalization (No Intervention): In this group, the former patients will experiment the standard of care, with an oncological follow-up.

INTERVENTIONS:
Other: Multidisciplinary day hospitalization — This multidisciplinary day hospitalization will consist at least of a psychological interview, an interview with a social worker and a medical interview. The objectives of this medical interview, conducted by a clinician researcher, are to summarize the pathology, the treatment(s) received, and to develop a personalized after-cancer plan.
  The psychological interview will assess the needs for further care, and will refer the former patient if necessary.
  The social interview will take stock of the former patient's return to school and/or professional life, and direct him/her to possible applications for social assistance if needed.
  If needs of supportive care emerge from the history of treatment period, some consultations can be added during the day hospitalization, like an interview with a dietician or an adapted physical activity assessment.
  Arms: Group A : former patients with multidisciplinary day hospitalization

SUMMARY:
Rational: 800 cases of cancer per year are diagnosed in France among Adolescents and Young Adults (AYA). This population has been specifically targeted since 2008 by the INCa, leading to the development of structures entirely dedicated to its management. Indeed, the occurrence of cancer in this period of transition leads to specific problems, which require a special attention. The various measures taken since then (Cancer Plan 2014-2019, DGOS instruction in 2016, 10-year strategy to fight cancer 2021-2030) have enabled the implementation of multidisciplinary structures, resulting in better access to care, and consideration of the social, family and relational dimensions of this population. However, the transition from the end of oncology treatment to the follow-up period remains a sensitive period, generating both positive (relief, joy) and negative feelings (uncertainty, feelings of abandonment, anxiety).

The investigators therefore hypothesize that the creation of a multidisciplinary end-of-treatment day hospital (DH) involving at least one medical interview, one psychological consultation and one social interview, would improve the quality of life of these former patients during the first year of oncology follow-up.

Method: This is a clinical research study conducted in a single centre. At their last visit for treatment, the study will be offered to patients. If the participants agree to participate, they will be randomized to benefit from DH in addition to their planned follow-up with their oncologist. The main objective is to compare the quality of life of former patients according to participation in DH or not. 210 patients will be included for a 20-month recruitment period.

Expected results: Throughout the development of DH, the investigators plan to improve the quality of life of former patients during this transitional phase.

DETAILED DESCRIPTION:
HOPAYA is a monocentric open-label clinical research with 2 parallel groups. Patients will be 1:1 randomly assigned in both groups.

The main objective of the study is to compare the evolution of the health-related quality of life of former patients who have benefited of a multidisciplinary day hospitalization to those who only had standard oncological follow-up during the first year after cancer treatment completion.

The secondary objectives are:

* to evaluate and compare the anxiety and depression level in both groups (with or without day hospitalization);
* to evaluate emotional competence in both groups (with or without day hospitalization);
* to evaluate the satisfaction about the multidisciplinary day hospitalization.

This study will be presented to patients (and their parents/legal tutors in case of minor patients) during the last visit for any treatment, by coordinating nurses of AYA Department and/or by the adult or pediatric oncologist. At the same time, the information sheet with the consent form will be provided in order to give them a reasonable time for reflection.

After the collection of the consent form for the conduct of the study, former patients will be randomly assigned in 2 groups, with or without multidisciplinary day hospitalization.

• Group A : former patients with multidisciplinary day hospitalization In this group, a multidisciplinary day hospitalization will be programmed after the end-of-treatment evaluation and 2 months after the end of treatment at the latest. This day hospitalization will consist at least of a psychological interview, an interview with a social worker and a medical interview. The medical interview will be conducted by a clinician researcher, specialised in long-term care after cancer. The objectives of this medical interview are to summarize the pathology, the treatment(s) received, and to develop a personalized after-cancer plan. The doctor will carry out both a clinical and an overall assessment of the patient, by wide-ranging questioning covering educational/professional, social, dietetic, addictology and physical fields. This medical interview is complementary to oncological follow-up, which consists of monitoring relapse and possible sequelae.

The psychological interview will be carried out if possible by the psychologist who followed the former patient during his/her treatment. The psychologist will assess the needs for further care, and will refer the former patient if necessary.

The social interview will be carried out by the social worker of AYA department. The social worker will take stock of the former patient's return to school and/or professional life, and direct him/her to possible applications for social assistance if needed.

If needs of supportive care emerge from the history of treatment period, some consultations can be added during the day hospitalization, like an interview with a dietician or an adapted physical activity assessment.

• Group B : former patients without multidisciplinary day hospitalization In this group, the former patients will experiment the standard of care, with an oncological follow-up.

The investigators expect that the AYAs' participation to the hospitalization day will positively impact their health-related quality of life compared to those who haven't participated. The investigators also expect that emotional competence will be explicative of the HRQoL through the mediation of the anxiety and depression levels.

Through the development of a multidisciplinary end-of-treatment day hospitalization, health care professionals plan to improve the quality of life of former patients during this transition phase of completing treatment. The lack of information on both medical and psychosocial long-term effects, will be improved by early and specific support. The feeling of abandonment often felt by former patients should decrease.

In addition, the early introduction of the long-term follow-up physician in the management of post-cancer, in parallel with the former patient's referring oncologist, should increase information and adherence to the personalized post-cancer plan.

The HOPAYA study aims to improve knowledge about the immediate quality of life after the treatment of AYAs with cancer, which is a challenge in this vulnerable population with specific needs. Comparison with the control group will make possible to highlight the specific impact of the establishment of a multidisciplinary end-of-treatment day hospitalization on quality of life. It will allow to target the flaws and shortcomings in AYA survivors support. The investigators also expect that the early screening of emotional competence will allow health care professionals to tailor support to the special needs of AYAs and their families.

Although many recommendations have emerged from the literature, to our knowledge, very few devices such this multidisciplinary day hospital have been elaborated for AYA early survivors of cancer. This study will evaluate the feasibility and the acceptability of a specific end-of-treatment hospitalization day for AYAs. The data collected and the analysed results in this study will allow to adapt and generalize this device in all AYAs' survivors in the CLB, and then at a larger level.

This study will lead to a scientific article published in an international journal, allowing the AYA hospitalization day to be reproduced in other oncologic centres and hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged between 15 and 25 years at diagnosis. This age range corresponds to the one chosen at the Leon Berard comprehensive cancer care center (CLB) for support in the AYA Department.
2. Be previously treated at the Paediatric Hematology and Oncology Institute (IHOPe) and/or at CLB in AYA Department
3. For a solid tumor or a lymphoma
4. Be in complete oncological response at the end of treatment; have received their end-of-treatment evaluation
5. Have finished their therapy since less than 2 months (therapy is defined by any treatment received, including maintenance)
6. Be capable of understanding, reading and writing French
7. Be affiliated to a health insurance plan
8. Have been informed of the study and have consented to it
9. For minor patients, consent of parents and/or legal tutors must be collected.

Exclusion Criteria:

1. cannot be followed-up throughout the duration of the study (12 months),
2. be deprived of liberty by a court or administrative decision,
3. have not consent to participate or are incapable of objecting in an informed manner.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 214 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Health-related Quality of life - emotional functioning | 12 to 15 months after cancer treatment completion
  The PedsQL is a standardised, generic assessment of health-related perceptions of quality of life in paediatric patients. The PedsQL consists of 4 subscale scores (physical, emotional, social and school) and 3 summary scores (physical health, psychosocial health and total scale). All PedsQL scores range from 0 to 100, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
To evaluate and compare the evolution of health-related quality of life at 12 months in the 2 groups | from 0 to 3 months after the end of the treatments, and at 12 months after cancer treatment completion
  The evolution of the QOL at 12 months will be studied via all the dimensions of QOL of the PedsQL questionnaire which will be completed by the patients of the two groups at inclusion ( from 0 to 3 months after the end of the treatments), and at 12 months
To evaluate and compare the evolution of QOL over time in the two groups: longitudinal analysis | at inclusion (0 to 3 months after the end of treatment), and at 3, 6, 9 and 12 months after cancer treatment completion
  The evolution of QoL will be measured via all the QoL dimensions of the PedsQL questionnaire which will be completed by patients in both groups at inclusion (0 to 3 months after the end of treatment), and at 3, 6, 9 and 12 months
To evaluate and compare the level of anxiety and depression in the 2 groups at inclusion (0 to 3 months after the end of treatment) and at 12 months | at inclusion (0 to 3 months after the end of treatment) and at 12 months after cancer treatment completion
  Anxiety and depression levels will be measured via the HADS questionnaire (Hospital Anxiety and Depression Scale) in the two groups (multidisciplinary DH in addition to standard oncology follow-up vs. standard oncology follow-up without multidisciplinary DH) at inclusion (0 to 3 months after the end of treatment) and at 12 months
To evaluate and compare the emotional regulation difficulties of the AYAs in the 2 groups at inclusion (0 to 3 months after the end of treatment) and at 12 months | at inclusion (0 to 3 months after the end of treatment) and at 12 months after cancer treatment completion
  Emotional regulation strategies will be measured using the DERS scale (Difficulties in Emotion Regulation Scale), in both groups (multidisciplinary DH in addition to standard oncological follow-up vs. standard oncological follow-up without multidisciplinary DH) at inclusion (0 to 3 months after the end of treatment) and at 12 months
To describe the compliance of the AJAs to the multidisciplinary DH vs. to the standard oncological follow-up without multidisciplinary DH, and to the proposed medical and paramedical orientations | 12 months after cancer treatment completion
  Compliance with follow-up will be described in the DH group by the number of DH proposed and actually performed (harvesting of the number of refusals and no-shows), as well as by the number and type of medical and paramedical consultations scheduled and actually performed in the two groups during the 12 months of follow-up
  * Group A: number of patients summoned to DH/number of DH carried out
  * Group A: oral reason for non-acceptance of the DH
  * Group A and B: number of patients called for the first oncology follow-up visit/number of visits made
  * Groups A and B: number and type of medical and paramedical consultations scheduled and actually performed during the 12 months of follow-up.
To describe the sequelae of the AJA in the 2 groups at inclusion (0 to 3 months after the end of treatment) and at 12 months | at inclusion (0 to 3 months after the end of treatment) and at 12 months after cancer treatment completion
  Sequelae will be described via the collection of clinical data carried out in the 2 groups (multidisciplinary DH in addition to the standard oncological follow-up vs. standard oncological follow-up without multidisciplinary DH) at inclusion (0 to 3 months after the end of treatment) and at 12 months
To evaluate the satisfaction of the AJAs who participate in the multidisciplinary DH following it | Immediately after the multidisciplinary DH
  Satisfaction with the DH will be assessed by means of a 10-point visual analogue scale completed by the AJAs following their participation in the DH

CONTACTS AND LOCATIONS:
Overall Officials: Amandine BERTRAND, MD, Principal Investigator — Institut d'Hématologie et d'Oncologie Pédiatrique
Locations (1):
- Centre Leon Berard, Lyon, France